CLINICAL TRIAL: NCT06051604
Title: A Prospective, Double-blind, Sham-controlled, Randomized Clinical Trial to Assess the Safety, Efficacy, Tolerability, and Optimal Dose of the Mi-Helper Device for Acute Treatment of Episodic Migraine in an at Home Setting.
Brief Title: Mi-Helper Transnasal Cooling for Acute Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CoolTech LLC (Industry)
Collaborators: ObvioHealth (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COT-001
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Episodic Migraine; Migraine With Aura; Migraine Without Aura; Migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding for this study will be applied to the Principal Investigator (PI) and the study team. The team members who are directly involved in the analysis of the study results, including the biostatistician, will also be blinded. Only the designated group of team members directly involved in overseeing the logistical and distribution aspects of the study products will be unblinded. As needed, the PI may be unblinded in case of an AE/SAE that may impact participant safety. If the unblinding occurs inadvertently or through PI's need due to an AE/SAE impacting participant safety, that event will be noted as a protocol deviation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Group I (sham) (Sham Comparator): 2 LPM of ambient air administered intermittently via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper
- Group II (active treatment 1) (Experimental): 4 LPM of dehumidified air administered via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper
- Group III (active treatment 2) (Experimental): 6 LPM of dehumidified air administered via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper
- Group IV (active treatment 3) (Experimental): 10 LPM of dehumidified air administered via Mi-Helper for 15 minutes
  Interventions: Device: Mi-Helper

INTERVENTIONS:
Device: Mi-Helper — The Mi-Helper device is a non-invasive, drug-free, novel therapy that uses a patented process of dry air flow across the nasal turbinates to induce a phase change (evaporation) that extracts energy (thermodynamics) causing local cooling which modulates nerves associated with pain and other symptoms of migraine. The device delivers a controlled pressure and flow of dry room temperature air along with a nebulized saline mist for added comfort and evaporative efficiency.
  Other Names: Mi-Helper transnasal cooling device

SUMMARY:
This is a prospective, double-blind, sham-controlled, randomized clinical trial . This study aims to assess the efficacy, safety, tolerability, and the optimal dose of the Mi-Helper transnasal cooling device for acute treatment of migraine in an at home setting.

Adults aged 18 years to 65 years old with a diagnosis of episodic migraine (with or without aura) for at least one year (self-reported) will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 65 years, inclusive of either sex at birth.
2. Lives in the contiguous United States.
3. Self-reported to be able to read and understand English sufficiently to provide informed consent.
4. Individual has had a diagnosis of episodic migraine with or without aura over at least 1 year, self-reported during screening.
5. Individual experiences 2 to 8 migraine attacks per month documented via migraine eDiary during screening.
6. Individual is in good reported general health at the time of screening.
7. Migraine onset before 50 years of age, self-reported during screening.
8. Migraine prophylaxis medication unchanged for 4 weeks prior to study enrollment.
9. Stated willingness to comply with all study procedures and availability for the duration of the study.
10. Individuals that own a functioning smartphone device, internet connection (Wi-Fi or data plan) and are willing to download the study app.

Exclusion Criteria:

1. Participant has difficulty distinguishing his or her migraine attacks from tension-type headaches.
2. Participant has 15 or more headache days per month reported via migraine eDiary and during screening.
3. Participant using any opioid medication at the time of screening.
4. Participant has received Botox treatment, barbiturates, supraorbital or occipital nerve blocks within the last 4 weeks of screening.
5. Participant lives at an altitude of 2000 meters or more above sea level.
6. Self-reported intolerance to intranasal therapy.
7. Self-reported recurrent epistaxis or chronic rhinosinusitis.
8. Self-reported sinus or intranasal surgery within the last 4 months of screening.
9. Self-reported history of 'complicated migraine or headaches' (i.e., hemiplegic migraine, ophthalmoplegic migraine, migrainous infarction, basilar migraine, post-traumatic headaches, post-concussion syndrome).
10. Known or suspected pregnancy as self-reported by the prospective participant at the time of screening.
11. Prospective participant unable to fully understand the consent process and provide informed consent due to either language barriers or mental capacity.
12. Self-reported diagnosis of alcohol or substance abuse disorder at the time of screening.
13. Participant with active chronic pain syndromes, such as fibromyalgia, chronic pelvic pain, or complex regional pain syndrome (CRPS); or other pain syndrome like trigeminal neuralgia.
14. Participant with severe psychiatric conditions (such as major depressive episode, bipolar disorder, major depressive disorder, schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
15. Failure to adhere to or inability to complete Study App inputs and onboarding activities during the screening period. Participants who are not adherent during the screening period are not eligible for study entry.
16. Prospective participant has participated in a migraine study or any interventional clinical study within the 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Pain relief at 2 hours post treatment | 2 hours
  From severe or moderate to mild or no pain, or from mild to no pain; based on the traditional 4-point VRS scale
Safety of the Mi-Helper device | 24 hours
  Measured by incidence of adverse events
Tolerability of the Mi-Helper device | 15 minutes
  Based on percent of participants who fail to complete the full treatment session

SECONDARY OUTCOMES:
Pain relief immediately post treatment | 0 minutes
  From severe or moderate to mild or no pain, or from mild to no pain; based on the traditional 4-point VRS scale
Pain relief at 24 hours post treatment | 24 hours
  From severe or moderate to mild or no pain, or from mild to no pain; based on the traditional 4-point VRS scale
Pain freedom immediately post treatment | 0 minutes
  A reduction of mild, moderate or severe pain at baseline to no pain.
Pain freedom at 2 hours post treatment | 2 hours
  A reduction of mild, moderate or severe pain at baseline to no pain.
Pain freedom at 24 hours post treatment | 24 hours
  A reduction of mild, moderate or severe pain at baseline to no pain.
Relief from most bothersome symptom (MBS) immediately post treatment | 0 minutes
  From severe or moderate to mild or none, or from mild to none; based on the traditional 4-point VRS scale
Relief from MBS at 2 hours post treatment | 2 hours
  From severe or moderate to mild or none, or from mild to none; based on the traditional 4-point VRS scale
Relief from MBS at 24 hours post treatment | 24 hours
  From severe or moderate to mild or none, or from mild to none; based on the traditional 4-point VRS scale
Freedom from MBS immediately post treatment | 0 minutes
  A reduction of mild, moderate or severe pain at baseline to none.
Freedom from MBS at 2 hours post treatment | 2 hours
  A reduction of mild, moderate or severe pain at baseline to none.
Freedom from MBS at 24 hours post treatment | 24 hours
  A reduction of mild, moderate or severe pain at baseline to none.

OTHER OUTCOMES:
Use of rescue medication 2-24 post treatment. | 24 hours
Participants belief of which treatment is received. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Parth Shah, MD, Principal Investigator — ObvioHealth
Locations (1):
- ObvioHealth, New York, New York, United States